CLINICAL TRIAL: NCT07111598
Title: Immunological Effects of Iron Supplementation in HHT Disease
Acronym: Fer&RO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL24_0724
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Haemorrhagic Telangiectasia
Keywords: Hereditary haemorrhagic telangiectasia (HHT); iron supplementation; lymphopenia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Lymphopenia

STUDY DESIGN:
Intervention Model Description: Patients will undergo the inclusion visit during a scheduled consultation at the HHT disease reference center in Lyon. Eligibility and exclusion criteria will be assessed at this visit by the principal investigator, based on blood test results obtained within 15 days prior to the consultation. In addition, six extra blood collection tubes will be drawn during the visit (D0), in addition to the routine blood samples., For patients in Groups 1 and 2, no follow-up visit will be scheduled. For patients in Group 3, iron supplementation will be administered as part of routine care within 14 days following inclusion, according to the patient's usual treatment protocol in terms of active compound, daily dosage, and treatment duration. A second consultation will be scheduled three months after inclusion (D+3 months) to assess the correction of iron deficiency and to collect six additional blood tubes for immunological analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No iron deficiency - no treatment (Experimental): Patients without iron deficiency with no need of iron supplementation. Ferritin > 25µg/L and no iron supplementation or red blood cell (RBC) transfusion over the past 3 months
  Interventions: Biological: Blood test at D0
- No iron deficiency under iron treatment (Experimental): Patient without iron deficiency thanks to iron supplementation or RBC transfusion Ferritin > 25µg/L and ongoing or recent (within the past 3 months) iron supplementation or RBC transfusion.
  Interventions: Biological: Blood test at D0
- Iron deficiency (Experimental): Patient with ferritin < 25µg/L No iron supplementation or RBC transfusion over the past 3 months
  Interventions: Biological: Blood test at D0; Biological: Blood test at D+3 months

INTERVENTIONS:
Biological: Blood test at D0 — Six extra blood collection tubes (28 mL) will be drawn during the visit (D0), in addition to the routine blood samples, at the blood collection center
Biological: Blood test at D+3 months — six extra blood collection tubes (28 mL) will be drawn during the visit (D+3 months) for group 3 patients, in addition to the routine blood samples, at the blood collection center
  Arms: Iron deficiency

SUMMARY:
Hereditary haemorrhagic telangiectasia (HHT), is a rare genetic vascular disorder with autosomal dominant inheritance. Its prevalence is estimated at approximately 1 in 6,000 individuals in France. Clinical manifestations include recurrent nosebleeds (epistaxis), cutaneous telangiectasias, and visceral arteriovenous malformations (AVMs) that may affect the lungs, gastrointestinal tract, liver, and brain.

Beyond vascular abnormalities, patients often present with a decrease in circulating T lymphocytes (T-cell lymphopenia), which can be profound but remains unexplained. There is also a distinct infectious risk profile associated with the disease: brain abscesses in the presence of pulmonary AVMs (pAVMs), and osteoarticular infections in patients with the longest durations of epistaxis. However, no definitive correlation has been established between T-cell lymphopenia and infection risk.

Iron-deficiency anemia is a frequent complication in HHT, affecting about 50% of patients, with a mean age of onset around 36 years. Its prevalence increases with age. These patients typically require prolonged and high-dose iron supplementation, administered either orally or intravenously, which may expose them to side effects not observed in other clinical contexts. In a previous study, we identified a correlation between the level of iron supplementation (none, oral, or intravenous) and the severity of T-cell lymphopenia.

This association may be explained by two potential mechanisms linking iron metabolism to immune function:

* A direct toxic effect of iron on immune system homeostasis
* Impaired lymphocyte production resulting from iron deficiency, with the type of supplementation serving as an indirect marker of deficiency severity We propose a prospective study designed to differentiate between these two hypotheses. The aim of the study is to characterize the impact of iron deficiency and iron supplementation on the immune system of patients with HHT.

ELIGIBILITY:
Inclusion Criteria:

* For all three groups:

  * Adult patient diagnosed with HHT (meeting 3 or 4 Curaçao criteria).
  * Documented pathogenic mutation in one of the following genes: ENG, ACVRL1, or MADH4.
  * Patient enrolled in the CIROCO cohort.
  * Written informed consent freely given and signed by the patient.
  * Patient covered by a social security scheme or equivalent.
  * Routine biological follow-up for HHT performed within the 15 days preceding the inclusion visit (complete blood count, reticulocytes, ferritin, CRP, calcium, phosphorus).
* Specific to Group 1:

  * Ferritin > 25 µg/L
  * No iron supplementation (oral or intravenous) in the past 3 months
  * No red blood cell transfusion in the past 3 months
* Specific to Group 2:

  * Ferritin > 25 µg/L
  * Ongoing oral iron therapy, or at least one intravenous iron infusion, or at least one red blood cell transfusion within the past 3 months
* Specific to Group 3:

  * Ferritin < 25 µg/L
  * No iron supplementation (oral or intravenous) in the past 3 months
  * No red blood cell transfusion in the past 3 months

Exclusion Criteria:

* Patients with hemoglobin levels < 90 g/L.
* Patients with active cancer or recent cancer remission (< 3 months) that may alter the immune profile.
* Patients with an active infection or recent infection recovery (< 3 months) that may alter the immune profile.
* Patients with an autoimmune or autoinflammatory disease, either active or recently treated (< 3 months), requiring immunosuppressive therapy and potentially altering the immune profile.
* Pregnant, postpartum, or breastfeeding women.
* Minors.
* Individuals deprived of liberty by judicial or administrative decision.
* Individuals undergoing psychiatric care.
* Individuals admitted to a healthcare or social institution for reasons other than research participation.
* Adults under legal protection (guardianship, curatorship).
* Individuals participating in another interventional clinical trial with an exclusion period still in effect at the time of pre-inclusion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Helper T-cell concentration (number of CD3⁺CD4⁺ lymphocytes per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.

SECONDARY OUTCOMES:
Naive/effector memory/terminal effector memory/central memory helper T lymphocytes concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.
Naive/effector memory/terminal effector memory/central memory cytotoxic T lymphocytes concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.
γδ T cells, mucosal-associated invariant T (MAIT) cells, and natural killer T (NKT) cells concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.
Natural killer (NK) cells concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.
Naive/memory/class-switched B lymphocytes concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.
Plasmablasts concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.
Classical/intermediate/non-classical/Tie2⁺ monocytes concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.
Myeloid and plasmacytoid dendritic cells concentration (number per mm^³ of blood). | Baseline for all the 3 groups and 3 months after iron supplementation for group 3.
  Samples will be analyzed by spectral cytometry to determine the concentration of each leukocyte population of interest.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No